CLINICAL TRIAL: NCT01722825
Title: Phase 1 Dose-Escalation Study of LY2157299 Monotherapy in Patients With Solid Tumors
Brief Title: Study of LY2157299 in Japanese Participants With Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14854; H9H-JE-JBAN (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-11-05; First posted 2012-11-07 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Neoplasms; Neoplasm Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — LY-2157299

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LY2157299 (Experimental): 80 up to 150 milligrams of LY2157299 administered orally, twice daily for 14 days, followed by 14 days with no study drug (2 weeks on/2 weeks off schedule) for at least two 28 day cycles. Participants receiving clinical benefit may continue receiving treatment until discontinuation criterion is met.
  Interventions: Drug: LY2157299

INTERVENTIONS:
Drug: LY2157299 — Administered orally.

SUMMARY:
The main purpose of this study is to evaluate the safety and side effects of LY2157299 in Japanese participants with advanced cancer or cancer that has spread to other parts of the body.

ELIGIBILITY:
Inclusion Criteria:

* Have histological or cytological evidence of a diagnosis of cancer that is advanced and/or metastatic. The participants must be, in the judgment of the investigator, an appropriate candidate for experimental therapy after available standard therapies have failed to provide clinical benefit for their disease.
* Have the presence of measurable or nonmeasurable disease as defined by the Response Evaluation Criteria in Solid Tumors.
* Have a performance status of higher than or equal to 1 on the Eastern Cooperative Oncology Group scale.
* Have adequate hematologic, hepatic and renal function.
* Have discontinued treatments for cancer excluding palliative treatments and recovered from the acute effects of therapy.
* Have discontinued treatment at least 28 days prior to the enrollment for an experimental agent that has not received regulatory approval for any indication.
* Are reliable and willing to make themselves available for the duration of the study and are willing to follow study procedures.
* Able to swallow tablets.
* Have an estimated life expectancy, in the judgment of the investigator, that will permit the participant to complete greater than or equal to 2 cycles of treatment.
* Males and females with reproductive potential: Must agree to use medically approved contraceptive precautions during the study and for 4 months following the last dose of study drug.
* Females with child bearing potential: Have had a negative urine/serum pregnancy test greater than or equal to 7 days before the first dose of study drug and must also not be breastfeeding. If female who stops breastfeeding enters the study, the female must stop breastfeeding from the day of the first study drug administration until at least 30 days after the last administration.

Exclusion Criteria:

* Have moderate or severe cardiac disease:

  * Have the presence of cardiac disease, including a myocardial infarction within 6 months prior to study entry, angina pectoris, New York Heart Association Class III/IV congestive heart failure, or uncontrolled severe hypertension.
  * Have documented major electrocardiogram abnormalities at the investigator's discretion.
  * Have major abnormalities documented by echocardiography with Doppler. Clinically non-significant abnormalities are excluded from this criterion.
  * Have persistently elevated brain natriuretic peptide or elevated Troponin I at screening local laboratory tests.
  * Have predisposing conditions that are consistent with development of aneurysms of the ascending aorta or aortic stress.
  * Have a history of cardiac or aortic surgery.
* Have current hematological malignancies.
* Have central nervous system metastases.
* Have serious preexisting medical conditions as follows;

  * Presence or history of interstitial pneumonitis
  * Uncontrollable severe diabetes
  * Presence of serious active infection or uncontrollable chronic infection
  * Presence of liver cirrhosis with Child-Pugh Stage of B or C
  * Other serious conditions judged by the investigator
* Have known positive test results in human immunodeficiency virus (HIV), hepatitis B surface antigen, or hepatitis C antibodies (HC Ab). Testing is not required unless circumstances warrant confirmation.
* In the opinion of the investigator or sponsor, are unsuitable for inclusion in the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2012-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Dose-Limiting Toxicities | Day 1 through Day 28 of Cycle 1

SECONDARY OUTCOMES:
Pharmacokinetics: Maximum Concentration (Cmax) of LY2157299 | Days 1, 3, 6 and 14 of Cycle 1 and Days 1 and 14 of Cycle 2
Pharmacokinetics: Area Under the Concentration-Time Curve (AUC) of LY2157299 | Predose up to 6 hours postdose on Days 1 and 14 of Cycles 1 and 2
Number of Participants with a Tumor Response | Baseline to study completion estimated at 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 ) or 1-317-615-4559 Mon - Fri 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559 ) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Tokyo, Japan

REFERENCES:
- [Derived] Fujiwara Y, Nokihara H, Yamada Y, Yamamoto N, Sunami K, Utsumi H, Asou H, TakahashI O, Ogasawara K, Gueorguieva I, Tamura T. Phase 1 study of galunisertib, a TGF-beta receptor I kinase inhibitor, in Japanese patients with advanced solid tumors. Cancer Chemother Pharmacol. 2015 Dec;76(6):1143-52. doi: 10.1007/s00280-015-2895-4. Epub 2015 Nov 3. PMID 26526984